CLINICAL TRIAL: NCT06511713
Title: Artificial Intelligence-Assisted Rapid Warning for Mental Disorders Based on High-Resolution Fundus Images and High-Speed Eye-Tracking Trajectories
Brief Title: AI-Assisted Rapid Warning for Mental Disorders Based on High-Resolution Fundus Imaging and High-Speed Eye-Tracking
Status: Recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Tianhong ZHANG, Professor, Shanghai Mental Health Center
Other Study IDs: SHDC2022CRD026
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Mental Disorder
Keywords: eye movement
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the Clinical High Risk for Psychosis (CHR) Group: Through the Structured Interview for Prodromal Syndromes/Scale of Prodromal Symptoms (SIPS/SOPS), the participants should meet the Criteria of Prodromal Syndrome. Participants should fulfill at least one of the prodromal syndrome criteria: (1) brief intermittent psychotic syndrome, (2) attenuated positive symptom syndrome, or (3) genetic risk and deterioration syndrome
  Interventions: Other: routine clinical treatment
- the Clinically Diagnosed Common Mental Disorders Group: 1,000 patients with common mental disorders, including 300 patients with schizophrenia, 300 patients with affective disorders, 200 patients with anxiety disorders, and 200 patients with cognitive impairment in the elderly.
  Interventions: Other: routine clinical treatment

INTERVENTIONS:
Other: routine clinical treatment — Participants will be informed that this is not a treatment study and it involves naturalistic follow-up without any extra intervention. They will otherwise follow the routine clinical treatment procedure.

SUMMARY:
This project aims to collect eye-tracking trajectories and fundus imaging data from individuals seeking mental health services. By utilizing artificial intelligence, combining dynamic (eye-tracking) and static (fundus) data, and employing convolutional neural network analysis methods, the investigators will develop models for the classification and early warning of common mental disorders. These models will assist clinicians in making objective diagnoses of common mental disorders and in predicting the risk of adverse outcomes, thereby addressing the significant technical bottleneck of the current lack of objective diagnostic and warning instruments for mental disorders.

DETAILED DESCRIPTION:
The investigators have completed the construction of the eye-tracking diagnostic and warning system and have piloted the new system. The plan is to recruit 1,000 individuals at Clinical High Risk for Psychosis (CHR) for model validation of predictive outcomes, and 1,000 patients with common mental disorders for model validation of diagnostic classification. This cohort includes 300 patients with schizophrenia, 300 patients with affective disorders, 200 patients with anxiety disorders, and 200 patients with cognitive impairment in the elderly. The system will also directly connect with the investigators' previous research data collection system and be deployed in no fewer than one hospital's healthcare system. Additionally, variables that may affect the accuracy of results will be fine-tuned to ensure that the eye-tracking and fundus system more accurately reflects actual clinical conditions. The application of the system will revolve around a big data analysis platform and seamlessly integrate with the existing hospital information systems, designing real-time feedback report modules to assist clinicians in making objective diagnoses efficiently and effectively.

ELIGIBILITY:
Inclusion Criteria:

* be aged 14 to 45-year-old
* have had at least 6-years of primary education
* be drug-naïve
* be understanding the survey, be willing to enrol in the study and sign the informed consent
* Through the Structured Interview for Prodromal Syndromes/Scale of Prodromal Symptoms (SIPS/SOPS), the participants should meet the Criteria of Prodromal Syndrome. Participants should fulfil at least one of the prodromal syndrome criteria: (1) brief intermittent psychotic syndrome, (2) attenuated positive symptom syndrome, or (3) genetic risk and deterioration syndrome
* Meets ICD-11 diagnostic criteria for schizophrenia
* Meets ICD-11 diagnostic criteria for mood disorders
* Meets ICD-11 diagnostic criteria for anxiety disorders
* Meets ICD-11 diagnostic criteria for neurocognitive disorders

Exclusion Criteria:

* Acute or chronic renal failure; liver cirrhosis or active liver diseases
* Abnormal laboratory tests results judged by the researchers to be clinically significant and considered to affect the efficacy of the test drugs or the safety of the subjects
* Severe or unstable physical diseases, including: neurological disorders (delirium, dementia, stroke, epilepsy, migraine, etc.), congestive heart failure, angina pectoris, myocardial infarction, arrhythmia, hypertension (including untreated or uncontrolled hypertension), malignant tumours, immune compromise, and blood glucose above 12 mmol/L
* Alcohol abuse within 30 days, or alcohol or drug dependence within 6 months before the trial
* Pregnant or lactating women, or women in childbearing age who are positive in urine human chorionic gonadotropin test, or men and women who do not take effective contraceptive measures or plan for pregnancy within 3 months after the initiation of the trial
* Stroke within the last month
* Participating in any clinical trial within 30 days before the baseline
* Other situations judged by the investigators not to be suitable for the clinical trial

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Help-seeking first-visit participants will be consecutively recruited from the Shanghai Psychotherapy and Psychological Counselling Centre at the Shanghai Mental Health Centre. They will be screened for eligibility by their clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Eye-tracking fixation point trajectory | 1 year
  Eye-tracking fixation point trajectory during free viewing of specific images by the participant (5 minutes)
Fundus examination | 1 year
  Color fundus imaging collected by a digital fundus camera (Canon CR-2) under non-mydriatic conditions of the participant

CONTACTS AND LOCATIONS:
Overall Officials: TianHong Zhang, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No